CLINICAL TRIAL: NCT03134261
Title: A Prospective Study Comparing the Diagnostic Accuracy of Bone SPECT-CT, Choline-PET-CT, PSMA-PET-CT, NaF-PET-CT and WB-MRI in the Detection of Prostate Cancer Bone Metastases
Brief Title: Diagnostic Imaging of Bone Metastases in Prostate Cancer Patients
Acronym: DIMAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Eva Dyrberg Mortensen, MD, Phd-student, Herlev Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DIMAB
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer Metastatic to Bone
MeSH Terms: interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Study participants will be allocated to the "ongoing project arm" at the time of enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPECT-CT (Other): The participants will undergo two project scans: WB-MRI and SPECT-CT
  Interventions: Diagnostic Test: WB-MRI; Diagnostic Test: SPECT-CT
- Cholin-PET-CT (Other): The participants will undergo two project scans: WB-MRI and Cholin-PET-CT
  Interventions: Diagnostic Test: WB-MRI; Diagnostic Test: Cholin-PET-CT
- PSMA-PET-CT (Other): The participants will undergo two project scans: WB-MRI and PSMA-PET-CT
  Interventions: Diagnostic Test: WB-MRI; Diagnostic Test: PSMA-PET-CT

INTERVENTIONS:
Diagnostic Test: WB-MRI — scanning methods
Diagnostic Test: SPECT-CT — scanning methods
  Arms: SPECT-CT
Diagnostic Test: Cholin-PET-CT — scanning methods
  Arms: Cholin-PET-CT
Diagnostic Test: PSMA-PET-CT
  Arms: PSMA-PET-CT

SUMMARY:
An improved diagnosis of bone metastases in prostate cancer patients can have a significant impact on treatment strategy and probably survival as well.

The primary purpose of the project is to determine the diagnostic accuracy of bone SPECT-CT, choline-PET-CT, PSMA-PET-CT, NaF-PET-CT and Whole-body MRI in the diagnosis of bone metastases in prostate cancer patients.

DETAILED DESCRIPTION:
The project is a prospective diagnostic test accuracy study. The project takes place at Herlev Hospital and is a collaboration between the Department of Radiology and the Department of Clinical Physiology and Nuclear Medicine.

The investigators want to include 300 prostate cancer patients referred to our standard diagnostic imaging (NaF-PET-CT scan) by the clinicians.

In addition to the standard diagnostic imaging (NaF-PET-CT-scan), two project will be performed on all participants. The project has three arms with the following scanning combinations:

A) Whole-body MRI + SPECT-CT B) Whole-body MRI + Cholin-PET-CT C) Whole-body MRI + PSMA-PET-CT The recruitment of project participants takes place on the day when the patients are undergoing a NaF-PET-CT scan in the course of regular clinical practice at our institution.

All readers are experienced radiologists or specialists in nuclear medicine. Patient identification on each scan will be anonymized and the reader will not have access to clinical and biochemical information or previous imaging studies.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for project participation if he meets all of the following criteria:

* Is either 1) a newly diagnosed prostate cancer patient in clinical suspicion of bone metastases or 2) a previously diagnosed prostate cancer patient in clinical suspicion of progression in the form of bone metastases. The subject must have been referred to the standard diagnostic imaging (18F-NaF-PET-CT) at our institution for bone metastases.
* The prostate cancer diagnosis must be biopsy-proven
* The subject is willing and able to comply with the protocol as judged by the investigator

Exclusion Criteria:

A subject will be excluded from the protocol if he meets one or more of the following criteria:

* Has prior malignancy, except for adequately treated basal cell or squamous cell skin cancer
* Has pacemaker or implanted devices (eg. cardiac valves, neurostimulator or insulin pump) that cannot be removed, metal clips/metal prostheses from surgery that are not MRI compatible or metallic foreign bodies in the eye (MRI exclusion criteria)
* Has any condition that places the subject at an unacceptable risk if he undergoes a diagnostic CT-scan (e.g. history of severe allergic reaction to the contrast agent).
* Has severe obesity (>195 kg is the weight limit for the scanner table)
* Has severe claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males can get prostate cancer
Enrollment: 300 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | The two project scans will be performed within a maximum of 30 days from the performance of the NaF-PET-CT scan
  Sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S. Thomsen, Professor, Study Director — Department of Radiology
Locations (1):
- Department of Radioogy/Department of Nuclear Medicine, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No